CLINICAL TRIAL: NCT02961400
Title: Improving Memory for Sleep Treatment Content With Text Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Allison Harvey, Professor of Clinical Psychology, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-02-4007_text_message
Record Dates: First submitted 2016-10-17; First posted 2016-11-11 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Sleep Wake Disorders
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Cognitive Behavioral Therapy; Chronotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PUSH text messages (Experimental): Participants will be sent text messages containing information relevant to their treatment condition (i.e., TranS-C or PE).
  Interventions: Other: PUSH text messages; Behavioral: TranS-C; Behavioral: PE
- PULL text messages (Experimental): Participants will be sent text messages containing information relevant to their treatment condition (i.e., TranS-C or PE). Text messages will request a response from the participant.
  Interventions: Other: PULL text messages; Behavioral: TranS-C; Behavioral: PE
- No text messages (Other): No text messages will be sent in this condition to participants in either treatment condition (i.e., TranS-C or PE).
  Interventions: Behavioral: TranS-C; Behavioral: PE

INTERVENTIONS:
Other: PUSH text messages — The intervention is designed to remind participants of treatment components.
  Arms: PUSH text messages
Other: PULL text messages — The intervention is designed to remind participants to recall treatment components.
  Arms: PULL text messages
Behavioral: TranS-C — The Transdiagnostic Sleep and Circadian Intervention (TranS-C) integrates evidence-based treatments derived from basic research on the circadian system.
  Other Names: Cognitive Behavior Therapy for Insomnia; Interpersonal and Social Rhythms Therapy; Chronotherapy
Behavioral: PE — Psychoeducation on the inter-associations between sleep, diet, exercise and stress.
  Other Names: Psychoeducation

SUMMARY:
A drop off in improvement over the months and years after treatment is common. One contributor may be poor memory for the contents of treatment. This study seeks to determine whether text messages containing reminders of the content of sessions will improve treatment outcomes.

DETAILED DESCRIPTION:
The growth in the use of technology provides an opportunity to send reminders to participants via text messages. The early studies on text messaging interventions indicate this approach is enjoyable for participants and has positive effects across a range of domains and treatment types. Hence, this study will test whether text messages containing reminders of the content of sessions will improve treatment outcomes. Two text messaging methods will also be tested. One is to send text messages to remind participants of their goals (PUSH condition) and the second is to send text messages to remind participants to recall their goals (PULL condition). This study will be conducted within the context of an NICHD-funded Randomized Controlled Trial (grant number R01-HD071065; protocol registration ID NCT01828320). In R01-HD071065 adolescents ages 10-18 (n = 176) will receive either the Transdiagnostic Sleep and Circadian Intervention (TranS-C) or a Psychoeducation (PE). At the 6-month follow-up assessment for R01-HD071065, participants will be randomized using 3 (PUSH text messages, PULL text messages, or no text messages) x 2 (TranS-C or PE) design. At the 6-month follow-up assessment, a questionnaire will also be administered to establish baseline memory for treatment. Participants will be sent text messages once per week until they return for the 12 month follow-up assessment for R01-HD071065. At the 12 month follow-up assessment, participants will be asked to complete the same memory for treatment questionnaire completed at the 6 month follow-up assessment as well as a questionnaire evaluating the acceptability of the text message reminders. This research is a first step toward identifying whether an inexpensive and ubiquitous technology (i.e., text messaging) can improve memory for treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Scoring within the lowest quartile of the Children's Morningness-Eveningness Preferences Scale (CMEP; 27 or lower) and a 7-day sleep diary showing a sleep onset time of of 10:40 pm or later for 10-13 year olds, 11 pm or later for 14-16 year olds, and 11:20 pm or later for 17-18 year olds at least 3 nights per week. Must have had the current pattern of late bedtimes for the last 3 months.
2. 'At risk' in one of the five health domains: emotional, behavioral, social, physical, and cognitive. Emotional risk will be operationalized as a score of 4 or above on any of the following items on the Child Depression Rating Scale: Difficulty Having Fun, Social Withdrawal, Irritability, Depressed Feelings, Excessive Weeping, or a T-score of 61 or above on the Multidimensional Anxiety Scale for Children (MASC), based on age group (10-11 years, 12-15 year, 16-19 years) using the MASC-10 Profile. Behavioral risk will be operationalized as a Sensation Seeking Scale score greater than 3.93 for males ages 10-13, greater than 3.19 for females 10-13, greater than 4.07 for males 14-18, or greater than 3.19 for females 14-18; taking ADHD medication or Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children (KSADs) diagnosis of ADHD; current alcohol or substance abuse; or past alcohol or substance dependence. Social and cognitive risk will be defined as "worse" than others the teen's age in one or more social behavior from Child Behavior Checklist (CBCL) Section VI or failing one or more academic class from CBCL Section VII, respectively. Physical risk will be operationalized as a Physical Health Questionnaire-15 score of 4 or above, six or more days of school absences, or a BMI above the 85th percentile for the participant's sex and age.
3. Age between 10 and 18 and living with a parent or guardian and and attending a class/job by 9am at least 3 days per week;
4. English language fluency;
5. Able and willing to give informed assent.

Exclusion Criteria:

1. An active, progressive physical illness (e.g., cancer, respiratory disorder) or neurological degenerative disease directly related to the onset and course of the sleep disturbance;
2. Evidence from clinical diagnosis or report by youth or parent of sleep apnea, restless legs or periodic limb movements during sleep. Youth presenting with provisional diagnoses of any of these disorders (e.g., sleep apnea) will be referred for a non-study polysomnography (PSG) evaluation at the parent's discretion and will be enrolled only if the diagnosis is disconfirmed;
3. Mental retardation, autism spectrum disorder, or other significantly impairing pervasive developmental disorder. Based on previous recruitment experiences in a youth depression study, it is expected that this exclusion will be invoked very infrequently (once every few years);
4. Bipolar disorder or schizophrenia or another current Axis I disorder if there is a significant risk of harm and/or decompensation if treatment of that comorbid condition is delayed as a function of participating in any stage of this study. Otherwise, all other comorbid psychiatric conditions will be allowed to (i) to maximize representativeness and (ii) because a byproduct may be that the treatment constitutes a helpful 'transdiagnostic' treatment for youth across psychiatric disorders.
5. A medication-free group may be difficult to recruit and would likely be unrepresentative. Hence, participants will not be excluded on the basis of stable use of medications (> 4 weeks). The exception was use of hypnotics and other medications known to alter sleep (e.g., melatonin).
6. History of substance dependence in the past six months;
7. Current suicide risk sufficient to preclude treatment on an outpatient basis.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 176 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Total sleep time (TST) average on weeknights via Daily Sleep Diary | Measured at 6-months post-treatment
  6mo TST
Total sleep time (TST) average on weeknights via Daily Sleep Diary | Measured at 12-months post-treatment
  12mo TST
Average bedtime on weeknights measured via Daily Sleep Diary | Measured at 6-months post-treatment
  6mo Avg Bedtime
Average bedtime on weeknights measured via Daily Sleep Diary | Measured at 12-months post-treatment
  12mo Avg Bedtime
Morning Eveningness preference measured via Childrens Morningness Eveningness Preference Scale | Measured at 6-months post-treatment
  6mo CME
Morning Eveningness preference measured via Childrens Morningness Eveningness Preference Scale | Measured at 12-months post-treatment
  12mo CME
Patient Recall of Session Contents | Change from 6-months post-treatment to 12-months post-treatment
  6-12mo Change in Patient Recall

SECONDARY OUTCOMES:
Sleepiness scale | Measured at 6-months post-treatment
  Embedded within the School Sleep Habits Survey
Sleepiness scale | Measured at 12-months post-treatment
  Embedded within the School Sleep Habits Survey
Pittsburgh Sleep Quality Index | Measured at 6-months post-treatment
  6mo PSQI
Pittsburgh Sleep Quality Index | Measured at 12-months post-treatment
  12mo PSQI
Discrepancy between weeknights and weekends for Total Sleep Time, Bedtime, and Waketime via Daily Sleep Diary | Measured at 6-months post-treatment
  6mo Weeknight-Weekend Differences
Discrepancy between weeknights and weekends for Total Sleep Time, Bedtime, and Waketime via Daily Sleep Diary | Measured at 12-months post-treatment
  12mo Weeknight-Weekend Differences
Text Message Evaluation | Measured at 12-months post-treatment
  Measure of the acceptability of receiving text messages
Child Behavior Checklist | Measured at 6-months post-treatment
  Parent measure
Child Behavior Checklist | Measured at 12-months post-treatment
  Parent measure

OTHER OUTCOMES:
Useful and Utilized Questionnaire | Measured at 6-months post-treatment
  6mo UUQ
Useful and Utilized Questionnaire | Measured at 12-months post-treatment
  12mo UUQ
Daily Sleep Diary | Measured at 6-months post-treatment
  total sleep time (weekend nights), weeknight bedtime, weekend risetime, total wake time (SOL+WASO) weeknights, total wake time (SOL+WASO) weekend nights, naps.
Daily Sleep Diary | Measured at 12-months post-treatment
  total sleep time (weekend nights), weeknight bedtime, weekend risetime, total wake time (SOL+WASO) weeknights, total wake time (SOL+WASO) weekend nights, naps.

CONTACTS AND LOCATIONS:
Overall Officials: Allison G Harvey, PhD, Principal Investigator — University of California, Berkeley; Michael R Dolsen, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States